CLINICAL TRIAL: NCT02533440
Title: A Prospective, Randomized, Open-Label Study Comparing Postsurgical Analgesia Using EXPAREL® To Standard Of Care For The Full Arch Surgical Therapy (FAST) Dental Implant Surgery Procedure
Brief Title: Efficacy of EXPAREL in Comparison to Standard of Care for the Treatment of Post Operative Dental Implant Pain
Acronym: FAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bellaire Facial Surgery Center (Other)
Responsible Party: Principal Investigator, Phillip T. Iero, Oral Surgeon, Bellaire Facial Surgery Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5142-001
Record Dates: First submitted 2015-08-12; First posted 2015-08-26 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthetics, Local; Analgesics, Opioid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EXPAREL and Local Anesthetics (Experimental): In the experimental group, patients will receive EXPAREL and local anesthetics, and will be prescribed opioid and non-opioid analgesics (for use only if in pain).
  Interventions: Procedure: EXPAREL and Local Anesthetics
- Oral Opioid and Local Anesthetics (Active Comparator): In the control group, patients will receive local anesthetics at the time of surgery and oral opioid or non-opioid analgesics (for use only if in pain).
  Interventions: Procedure: Oral Opioid and Local Anesthetics

INTERVENTIONS:
Procedure: EXPAREL and Local Anesthetics — Patients will receive EXPAREL and local anesthetics, as well as opioid and non-opioid analgesics prescription, (only use if needed, for post surgical pain)
  Arms: EXPAREL and Local Anesthetics
Procedure: Oral Opioid and Local Anesthetics — Patients will receive local anesthetics, as well as oral opioid or non-opioid analgesics, (only use if needed, for post surgical pain)
  Arms: Oral Opioid and Local Anesthetics

SUMMARY:
This study is researching managing postsurgical pain by injecting both short-acting local anesthetics and EXPAREL® at the time of surgery and reviewing if it could reduce or eliminate the need for postsurgical opioids and improve clinical outcomes following the FAST dental implant surgery procedure. This approach is being compared to the current standard of care.

DETAILED DESCRIPTION:
Postsurgical pain following the Full Arch Surgical Therapy (FAST) dental implant surgery procedure is commonly managed with a variety of interventions, including local infiltration with short-acting local anesthetics during surgery and the use of postsurgical opioid and non-opioid analgesics. Although this approach to managing postsurgical pain is considered the current standard of care, its reliance on opioid analgesics to provide analgesia beyond the duration of short-acting local anesthetics exposes patients to opioid-related adverse events (ORAEs) that may delay their recovery and have other deleterious clinical consequences. The primary objective of this study is to determine the efficacy and safety of local infiltration of EXPAREL for the FAST dental implant surgery procedure compared to standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older;
* Ability to speak, read, and write in English;
* Ability to communicate via telephone;
* Scheduled to undergo FAST dental implant surgery procedure at a study center within the next 30 days for both maxillary and mandibular repair with at least 4 upper and 4 lower teeth to be extracted;
* Willing to provide informed consent, participate in study, and comply with study protocol.

Exclusion Criteria:

* Daily opioid consumption for more than 30 days prior to surgery;
* Any opioid consumption within 3 days prior to surgery.
* Prior treatment for alcohol, recreational drug, or opioid abuse.
* Hypersensitivity or allergy to local anesthetics, non steroidal anti-inflammatory drugs, or opioids;
* Breastfeeding, pregnant, or contemplating pregnancy prior to surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2015-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Postsurgical Pain Severity | 7 days

SECONDARY OUTCOMES:
Food ingesting tolerance | 7 days
  Ability to ingest different foods
Analgesic medication use | 7 days
  Analgesic medication use
Patient Satisfaction | 7 days
  Patient Satisfaction with pain control
Incidence of ORAEs and other adverse events (AEs) | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Phil Iero, M.D., DDS, Principal Investigator — Primary Investigator
Locations (3):
- United States (3):
  - ClearChoice Dental Implants, Atlanta, Georgia
  - ClearChoice Dental Implants, Houston, Texas
  - ClearChoice Dental Implants, The Woodlands, Texas